CLINICAL TRIAL: NCT03677661
Title: Cervico-vestibular Rehabilitation for Mild Traumatic Brain Injury - A Randomized Clinical Trial
Brief Title: Cervico-vestibular Rehabilitation for Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale (Other); Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Pierre Langevin, Professeur de Clinique, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Quebec mTBI
Record Dates: First submitted 2018-09-15; First posted 2018-09-19 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Post-Concussion Syndrome; Mild Traumatic Brain Injury; Vestibular Disorder; Whiplash Injuries; Concussion, Brain
Keywords: Concussion; Physical therapy; Vestibular rehabilitation; Mild traumatic brain injury
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion; Vestibular Diseases; Whiplash Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional approach (Active Comparator): Graded aerobic exercise and advice for graded cognitive stimulation approach based on the 2016 Berlin consensus
  Interventions: Other: Conventional approach
- Personalized rehabilitation program (Experimental): Cervico-vestibular rehabilitation personalized patient-centered clinical program combined with the exercise and advice of the conventional approach
  Interventions: Other: Personalized rehabilitation program

INTERVENTIONS:
Other: Conventional approach — The intervention will consist of light cognitive and physical activity with no symptoms exacerbation followed by graded exertion. Participant will be evaluated by a neuropsychologist. The neuropsychological intervention will consist of advice relative to cognitive rest in line with the clinical evaluation results followed by an individualized step-by-step graded exposition to cognitive stimulus according to symptoms evolution. A kinesiologist will also evaluate the symptoms response to cardio-vascular exertion. According to the result of this clinical evaluation, a graded physical exercise program will be given to the participants. 8 in-clinic cardio-vascular exercise sessions in a 6-week period supervised by the kinesiologist (30 to 45 minutes each session) will be provided.
  Arms: Conventional approach
Other: Personalized rehabilitation program — The same advice and exercise program than the active comparator group will be provided. However, 2 physiotherapists will provide 8 treatment session ( 30 to 45 minutes). One physiotherapist will initially evaluate the physical dysfunctions associated to mTBI with a standardized evaluation to build the treatment plan. He will provide cervical manual therapy and therapeutic exercises based on the best current clinical approach and according to the impairment specifically found initially. A vestibular physiotherapist will provide treatment of canalith repositioning manoeuvre, vestibular adaptation, ocular motor exercises, balance and/or habituation exercises. This treatment will be adapted to the individual patient. No more than 8 sessions will be delivered.
  Arms: Personalized rehabilitation program

SUMMARY:
Neck pain, dizziness and headache are common symptoms following mild traumatic brain injury (mTBI). The efficacy of cervical spine and vestibular-ocular system impairments intervention need to be determined. In this randomized clinical trial, a 6-week personalized clinical rehabilitation program on subacute mTBI will be compare to a conventional approach. The rehabilitation program will include cervical spine exercise combined with manual therapy as well as vestibular-ocular rehabilitation. Overall symptoms will be measured by the Post-Concussion Symptoms Scale (PCSS). Disability and symptoms severity related with neck pain, headache and dizziness will also be evaluated after the treatment period and at 6-week post-treatment.

DETAILED DESCRIPTION:
BACKGROUND

Mild traumatic brain injury (mTBI) is an acknowledged public health problem. It is estimated that between 1.6 to 3.8 million brain injuries occur annually in the United States, with up to 75% classified as mild. The majority of mTBI resolves within 10 to 14 days. However, up to 31% of pediatric cases and 25% of adult cases present post concussive syndrome (PCS), which is a persistence of somatic (for example: headache, neck pain, dizziness, nausea, balance dysfunction), cognitive (for example: memory loss and slowed reaction time), and/or psychological (for example: depression and anxiety) symptoms. Among these symptoms, headache and dizziness are the most commonly reported, followed by nausea and neck pain. Many of these PCS symptoms could be explained by injuries to structures near or in the head, other than the brain itself. For example, following a trauma, structures such as the cervical spine, the vestibular ocular system and the temporomandibular joint can be injured. The energy needed to produce an mTBI can be transferred to the neck and produce an injury mechanism similar to the one observed in whiplash associated disorders (WAD). Neck pain, headaches, dizziness and balance dysfunction are common symptoms associated with both mTBI and WAD. Specific interventions for these injuries are therefore needed when present.

For individuals presenting persistent post-concussion symptoms, the most recent international consensus statement (2017 Berlin consensus on concussion in sport) recommends the addition of an individualized rehabilitation approach to the usual rest and sub-symptoms gradual activation strategies. However, this new recommendation is based on weak evidence as well as expert recommendations. Therefore, the effects of adding individualized rehabilitation interventions for the treatment of potential impairments of body function associated with neck pain, headache and dizziness, needs to be evaluated in individuals with mTBI. The treatment of neck pain, cervicogenic headache, dizziness and balance dysfunction with multimodal rehabilitation interventions or vestibular rehabilitation has been demonstrated effective in several systematic and Cochrane reviews; however none of the randomized control trials (RCT) included in these reviews included individuals with mTBI. Two RCTs have partially looked at the effects of rehabilitation interventions in some subgroups of mTBI patients. One RCT (n=31) has demonstrated that patients with sport-related concussion treated with a standardized combination of vestibular and cervical physiotherapy were quicker to be medically cleared to return to sport than a control group who was resting and gradually returning to activities. However, the intervention used in that study was not individualized to the specific impairments of the participants. Another RCT recruited 41 sport-related concussion patients with dizziness as the main symptom and found that a rehabilitation treatment targeting dizziness was more effective in terms of time to medical clearance than a minimal intervention (subtherapeutic and non-progressive therapeutic techniques). However, as a most likely multifactorial condition, mTBI treatments arguably need to be individualized to the patient's clinical presentation and the outcomes need to encompass all types of symptoms. In that context, there is a need for further RCTs evaluating the effect of a personalized patient-centered rehabilitation approach (based on the Berlin consensus) on mTBI.

Objectives and hypothesis: The primary objective of the current RCT is to compare the addition of a 6-week personalized patient-centered clinical rehabilitation program to a conventional approach in adults with subacute (> than 3 weeks post TBI) headache, neck pain and /or dizziness-related to mTBI on the severity and impact of symptoms as measured by the Post-Concussion Symptoms Scale (PCSS). The secondary outcomes will be: clearance to return to usual activities, number of recurrence episode, functional level, neck pain, headache and dizziness. Our hypothesis is that the personalized patient-centered clinical rehabilitation program will improve overall symptoms, time to return to activities as well as function faster than the conventional approach and between group differences will be observed at week 6, 12 and 26.

METHODS

Study Design: This single-blind, parallel-group RCT will include 8 supervised treatments during a 6-week rehabilitation program (2 sessions/week the first 2 weeks, then 1 session/week for the last 4 week) and four evaluation sessions over 26 weeks (baseline, week 6 [immediately after the rehabilitation program], week 12 [6 week after the end of the rehabilitation program] and week 26). All participants will take part in the baseline evaluation. After giving an informed consent, they will first complete a questionnaire on sociodemographic (age, gender, type of sport or physical activities, number of years playing sport and/or other activities), symptomatology (mechanism of injury, history of previous mTBI, history of dizziness, headache, neck pain and unsteadiness) and comorbidity, as well as self-administered questionnaires that evaluate symptoms and functional limitations, including the PCSS (primary outcome). Once baseline data collected, participants will be randomly assigned to the control or intervention group. The control group will receive a the 6-week conventional intervention based on sub-symptoms gradual cardio-vascular exercise program. The experimental group will receive a 6-week personalized patient-centered clinical rehabilitation program in addition to the same intervention as the control group. Between week 6 and week 12, participants will be asked to continue their exercises and follow the advice given at the last meeting with the health professional. Six, 12 and 26 weeks after randomization, all the outcomes will be revaluated. The evaluation sessions will be carried out at the Centre interdisciplinaire de recherche en réadaptation et en intégration sociale (CIRRIS) by a research assistant blinded to group assignment, while the interventions will be given at Clinique Cortex by experienced physiotherapists, neuropsychologists and kinesiologists.

Population: 46 adults presenting to the Clinique Cortex (Concussion clinic) with a diagnosis of mTBI (based on the definition of the Berlin 2016 international consensus statement) and persistent symptoms of dizziness, neck pain and/or headaches (reported on the PCSS)17 lasting for more than 3 weeks will be recruited. The reported symptoms must 1) have started in the first 72 hours following an impact, 2) include one or more cognitive symptom(s), as found in the PCSS).

Sample size calculation is based on changes evidenced by the PCSS for individuals with mTBI. According to sample size calculation (G*Power 3.1.9.2; α=0.05, effect size=0.8, power [1-β]=0.80, Standard Deviation(SD)=20.0 PCSS points, Minimal Detectable Change (MDC)=12.3 PCSS points, 10% attrition), a minimum of 23 patients are needed in each group. Therefore, 46 participants with mTBI will be recruited.

Inclusion and exclusion criteria are described elsewhere in the form.

Randomisation/Blinding: A randomisation list will be generated by an independent research assistant (not involved in data collection) prior to the initiation of the study using a random number generator. Allocation will be concealed in sealed and opaque envelopes that will be sequentially numbered. A blocked randomisation will be used to make sure that two equal groups of 23 participants are obtained. Stratification will be done according to sex to ensure women and men are equally represented in each group as it has been shown that women tend to recover more slowly than man from a mTBI. Given that it is not possible to blind the treating physiotherapist and the participants, a single-blind design will be used as only the evaluator will be blinded. One of the Principal Investigator (PI) will open the randomisation envelope indicating the participant's assignment and will send the information to the treating therapist. The physiotherapists, neuropsychologists and the kinesiologists will be blinded to the baseline evaluation results. To evaluate the effectiveness of blinding, the evaluator will complete a question related to her/his opinion of the allocation. Participants will be unaware of the treatment provided to other participants. Participants will be instructed not to reveal or discuss treatment with the evaluator. To assess blinding effectiveness, the evaluator will answer the following question at the week-6 evaluation: "In your opinion, which intervention this participant received?" The possible answers are: 1) conventional (comparison group); 2) intervention testing the personalized patient-centered clinical rehabilitation program (experimental group); 3) I have no idea.

The outcome measures are well described elsewhere in the form.

Statistical Analyses: Descriptive statistics will be used for all outcome measures at each measurement time to summarize results. Baseline demographic data will be compared (independent t-test and Chi-squared tests) to establish the comparability of groups. All data will be tested to check the distributional assumptions for the inferential statistical analyses. An intention-to-treat analysis will be used in which all participants will be analysed in the group to which they were originally assigned. Per protocol analysis will also be performed. All dropouts and the reason for dropping out of the study will be reported. Any harm or unintended effects during the programs will be recorded. A 2-way ANOVA (2 Groups [Group 1 or 2] x 4 Time [week 0, 6, 12, 26]) will be used to analyse the effects of the rehabilitation programs on the primary outcome and on most of the secondary outcomes (SPSS 22, proc GENLIN). We expect no group effects, as the groups should be equal at baseline. A time effect should be observed, as both groups should improve given they will both receive an interventions. Finally, we expect a significant Time x Group interaction since the groups should react differently over time, with a faster recovery for the Experimental group seen at week 6 and 12. This will be statistically detailed with post-hoc tests (Bonferroni correction). An independent t-test will be used to analyse the effects of the rehabilitation programs on clearance to return to function.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age;
* Sustained a mTBI in the past 3 to 12 weeks;
* Having ongoing post-concussion symptoms from the list in the PCSS that started 72 hours or less after an impact;
* Having felt at least one or more cognitive symptoms that started 72 hours or less after an impact;
* Having abnormalities on one of the following test : the cervical physical examination (eg, tenderness/spasm on segmental testing, or reduced motion), the vestibular evaluation (eg, Dix hallpike test, vestibulo-ocular reflex test, or head thrust test) or the ocular motor evaluation (eg, convergence, smooth visual pursuits, or saccades).

Exclusion Criteria:

* Patients with more than 30 minutes of loss of consciousness for the current episode;
* Patients with more than 24 hours of post-traumatic amnesia;
* Glasgow Coma Scale score lower than 14 at the time of injury;
* Patients with radiographic evidence of subdural hemorrhage, epidural hemorrhage, intraparenchymal hemorrhage, and cerebral or cerebellar contusion;
* Post-injury hospitalization for more than 48 hours;
* Fracture (head, neck and spine);
* Having a neurological condition, other than the actual mTBI;
* Having a cognitive or behavioural impairment with participation in the study;
* Have had general anesthesia during the three-month period prior to the study;
* Having received physiotherapy tretament for the currwnt episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Post-Concussion Symptoms Scale (PCSS) | 26 weeks post-intervention
  The severity and impact of symptoms will be measured by a self-reported scale, the PCSS. This scale is a list of 22 symptoms for which participant rate each symptom for severity on a 0 (none) to 6 (severe) numerical scale. The maximum possible score is 132 (22 x 6 = 132). This valid and reliable scale has a minimal detectable change (90% confidence interval) of 12.3 PCSS points. Normative values have been established. The symptoms list can be divided in four main sub-groups (physical, cognitive, emotional and sleep disorders) and analysed accordingly.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 26 week post-intervention
  The level of neck pain and headache will be captured separately with NPRS. Using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable), participants will be asked to answer the following question: "On a scale of 0 to 10, where 0 corresponds to no pain and 10 to the worst imaginable pain, evaluate the intensity of your neck pain at this moment". The same question will be asked for the headache. The NPRS is moderately reliable (ICC = 0.76) and has a clinically important difference of 13%.
Neck Disability Index (NDI) | 26 week post-intervention
  The NDI is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. Questions include pain and activities of daily living. The questions are measured on a six-point scale from 0 (no disability) to 5 (full disability). The numeric response for each item is summed for a total score ranging from 0 to 50. The reliability (Intraclass Correlation Coefficient [ICC]: 0.73 to 0.98), construct validity, and responsiveness to change have all been demonstrated in various populations. The validated French version NDI will be used.
Headache Disability Inventory (HDI) | 26 week post-intervention
  The HDI is a 25-item questionnaire measuring the disability related to patient reported headache. Questions include activities of daily living and perceived disability as measured with an ordinal scale (yes (4 points), sometimes (2 points), no (0 point)). After adding every numerical score, the total score is on 100 for which 0 means no disability and 100 complete disability. The test-retest reliability (r=0,79 to 0,83) and the minimal detectable change (16 points) are known.
Dizziness Handicap Inventory (DHI) | 26 week post-intervention
  The DHI is a 25-items questionnaire. The items are sub grouped into three content domains representing functional, emotional, and physical aspects of dizziness and unsteadiness. The purpose of this scale is to identify difficulties that the patient may be experiencing because of dizziness or unsteadiness. The questionnaire demonstrated high Test-retest reliability (r = 0.92 to 0.97) and internal consistency (α = 0.72 to 0.89).
Global Rating of Change | 26 week post intervention
  GRC questions are designed to quantify a patient's perceived improvement or deterioration over time. Using a 15-point GRC scale, ranging from -7 (a very great deal worse) to 0 (about the same) to +7 (a very great deal better), participants will be asked to answer the following question: " Overall, has there been any change in your condition since the initial evaluation? Please indicate if there has been any change in your condition by choosing one of the following options." The validity, reliability (ICC = 0.90) and responsiveness of GRC scales have been established.
Cervical flexion rotation test | 12 week post intervention
  The inter-examiner reliability (ICC = 0.87 - 0.96) and validity to diagnose cervicogenic headache (positive likelihood ratios from 5 to 10) of the FRT are known. The test result is presented as a right-left rotation difference. A difference of more than 10 degrees is a cervicogenic headache diagnostic criterion.
Vestibular/Ocular Motor Screening (VOMS) | 12 week post intervention
  The VOMS has a good internal consistency (α = 0.97) and reliability (ICC = 0.89 - 0.98). It consisted of 5 tests: visual pursuit, visual saccade, near point convergence, vestibulo-ocular reflexes (horizontal and vertical), and visual motion sensitivity test. The numerical rating scale of symptoms increasing is recorded for each test (0 to 10 scale (0=better, 10=worse). For the near point convergence 3 measures are taken and a mean of those measure is calculated. Each of the 5 tests are reported separately.
Head impulse test | 12 week post intervention
  This test evaluates whether the eyes gaze can stay still in front by looking at a target when the head is rapidly rotated to the right or the left at a small amplitude (5-10 degrees) by the evaluator. The test is considered positive when a corrective saccade is observed immediately after the rotation of the head. The specificity (82%) and sensitivity (71 to 84%) are known to determine a bilateral or unilateral vestibular hypofunction.
Recurrence episodes | 26 week post-intervention
  number of recurrence episodes calculated as the number of episodes of symptoms with a duration of at least 48 hours following a trauma during the 26 weeks of the study
Clearance to return to function | immediately post-intervention
  The number of days between the initial evaluation and the full clearance to return to function will be measured. The clearance to return to function will be determined by the treating therapist and the neuropsychologist. The treating therapist will use the stepwise progression of the 5th International Consensus Statement on Sport Concussion. When the patient will achieve the last step of this progression which means that the patient can safely return to play, the neuropsychologist and the kinesiologist will confirm the decision with a structured interview (neuropsychologist) and an aerobic test (kinesiologist). The clearance will be determined by the day for which 1) the symptoms will have resolved 2) the neurological, cervical spine and vestibular exams will be deemed normal by the treating physiotherapist 3) the subject returned to his normal level of all functional activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, pht, PhD, Study Director — Professor; Pierre Frémont, MD PhD, Study Director — Professor
Locations (1):
- Clinique Cortex, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
On demand directly to research team
Supporting Information: Study Protocol, CSR
Time Frame: Available
Access Criteria: https://pubmed.ncbi.nlm.nih.gov/31737275/ https://pubmed.ncbi.nlm.nih.gov/35102743/
URL: https://pubmed.ncbi.nlm.nih.gov/31737275/

REFERENCES:
- [Derived] Langevin P, Fremont P, Fait P, Dube MO, Roy JS. Moving from the clinic to telehealth during the COVID-19 pandemic - a pilot clinical trial comparing in-clinic rehabilitation versus telerehabilitation for persisting symptoms following a mild Traumatic brain injury. Disabil Rehabil. 2024 Jun;46(13):2880-2889. doi: 10.1080/09638288.2023.2236016. Epub 2023 Jul 19. PMID 37466379
- [Derived] Langevin P, Fait P, Fremont P, Roy JS. Cervicovestibular rehabilitation in adult with mild traumatic brain injury: a randomised controlled trial protocol. BMC Sports Sci Med Rehabil. 2019 Nov 11;11:25. doi: 10.1186/s13102-019-0139-3. eCollection 2019. PMID 31737275